CLINICAL TRIAL: NCT04048733
Title: Timely Acquirement of 12-lead Electrocardiography Using Patchy-type Wireless Device Among Patient With Chest Pain in Emergency Departement
Brief Title: Timely Acquirement of 12-lead ECG Using Patchy-type Wireless Device Among Patient With Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-01-046
Record Dates: First submitted 2019-07-31; First posted 2019-08-07 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Chest Pain; Electrocardiography
Keywords: Electrocardiography; Chest pain; Emergency Service,Hospital; Wireless Technology
MeSH Terms: conditions — Chest Pain; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patchy type-lead ECG (Experimental): ED physicians will prescribe to perform second and third 12-lead ECG in every 15 minutes.
  Second and third 12 lead ECG will be taken using patchy-type 12-lead ECG device as a doctor's order. This device will be automatically record 12-lead ECG 3 times in 1 minutes at a time by its algorithm.
  Interventions: Device: patchy-type wireless 12-lead ECG
- Standard 12-lead ECG (No Intervention): ED physicians will prescribe to perform second and third 12-lead ECG in every 15 minutes.
  Second and third 12 lead ECG will be taken using standard 12-lead ECG device as a doctor's order. Interns and ECG technicians will perform 12-lead ECG as they perform as usual.

INTERVENTIONS:
Device: patchy-type wireless 12-lead ECG — Perform 12-lead ECG using patchy-type wireless 12-lead ECG. This device automatically record 12-lead ECG in every 15 minutes by its algorithm.
  Arms: Patchy type-lead ECG

SUMMARY:
In this study, the investigators compare timely acquirement of 12-lead ECG using patchy-type wireless versus using standard 12-lead ECG system among patient with chest pain in ED. The purpose of this study is to determine the difference of timely acquirement of 12-lead ECG using two different systems and the difference of hospital delay in ED between two groups. The participants were randomly divided into 2 groups: one performing an ECG examination using the standard 12-lead ECG and the other using the patch-type mobile 12-lead ECG.The 12-lead ECG will be taken 2 times serially in every 15 minutes.

DETAILED DESCRIPTION:
1. research background Electrocardiography (ECG) is the most important diagnostic tool for rapid detection of acute coronary syndrome, and should be performed and interpreted promptly on appearance of symptoms. Early detection of ST-elevation myocardial infarction (STEMI) on a 12-lead ECG, within 10 minutes after the first medical contact before hospitalization not only minimizes the time taken for diagnosis and reperfusion therapy but also increases the chances of patient survival and preservation of myocardial function.

   However, it is challenging to perform a 12-lead ECG promptly using the standard 12-lead ECG system for several reasons. First, it is difficult to identify the landmarks for the 10-electrode configuration of the standard ECG. Second, electrodes on the extremities often cause artifacts due to body and muscle movements. Moreover, most of the standard 12-lead ECG systems have cables connected to the precordial and limb leads, which frequently get entangled and disorganized, and can be difficult to manage.Most importantly, its accuracy is dependent on the operators' experience; not just that of the nurses or emergency medical technicians, but also of cardiologists.These difficulties might increase the time taken to perform an ECG especially in pre-hospital situations.
2. Objective The purpose of this study is to determine the difference of timely acquirement of 12-lead ECG using two different systems and the difference of hospital delay in ED between two groups.
3. Design : Randomized controlled trial
4. Setting : ED at the Samsung medical center
5. Enrollment : 36 patients who visited the ED with chest pain
6. Intervention Standard 12-lead ECG will be performed at the time of visiting ED to the participants with chest pain.

ED physicians will prescribe to perform second and third 12-lead ECG in every 15 minutes.

1. Control group : Second and third 12 lead ECG will be taken using standard 12-lead ECG device as a doctor's order.
2. Study group :Second and third 12 lead ECG will be taken using patchy-type 12-lead ECG device as a doctor's order.

7. scoring To measure, interval from the anticipated time to take 12-lead ECG to the time actually performed will be measured. The duration from the anticipated time to the time of verification by physician will be also measured.

8. study period The experiment ends when patient who agreed to participate in the study discharged the ED.

ELIGIBILITY:
Inclusion Criteria:

* A subject who visited the ER with a cardiogenic chest pain
* adult patients over 19 years of age
* A subject who completed the 1st ECG

Exclusion Criteria:

* A subject who did not agree with this study
* arrest patient
* Dead on arrival
* STEMI patients who confirmed by 1st ECG in ER
* shock status patient in triage state

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Time from ordering to performing 12-lead ECGs during up to 24 hours in ED. | measure the time duration from ECG ordering to performing during up to 24 hours in ED
  Comparison of interval from the anticipated time to take 12-lead ECG to the time actually performed will be measured.
Time from ordering to verifying 12-lead ECGs by ED physician during up to 24 hours in ED. | measure the time duration from ECG ordering to verifying by ED physician during up to 24 hours in ED
  Comparison of interval from the anticipated time to take 12-lead ECG to the time verified by physician

SECONDARY OUTCOMES:
The Presence of artifacts in 12-lead ECGs. | ECG reading and checking of presence of artifacts in 12 lead ECGs through study completion, an average of 1 month.
  Comparison of the presence of artifacts in 12-lead ECGs in intervention group and control group

CONTACTS AND LOCATIONS:
Overall Officials: wonchul cha, doctoral, Principal Investigator — samsumg medical center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: No